CLINICAL TRIAL: NCT04762173
Title: Self-Help for Stress Related to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Michelle G. Newman, Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015766
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Stress
Keywords: Self-help; Internet; Cognitive-behavioral therapy; Positive psychology; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online self-help intervention (Experimental): Participants are provided access to two online self-help programs provided by SilverCloud Health. One program is designed to support general stress resilience using principles and techniques from positive psychology and cognitive-behavioral therapy. The other program is designed to support coping with pandemic-related stressors using psychoeducation and cognitive-behavioral therapy and grief therapy principles. Participants have access to both programs and can proceed through them in the order and pace of their choosing. The online self-help intervention is fully self-guided.
  Interventions: Device: Online self-help intervention
- Care as usual (No Intervention): Participants are provided information about how to contact the counseling center at their college and/or in the local community using the phone number and website of their counseling center (if available), as well as the Substance Abuse and Mental Health Services Administration treatment locator.

INTERVENTIONS:
Device: Online self-help intervention — Access to two online, self-guided programs available on the SilverCloud Health website.
  Other Names: SilverCloud Health
  Arms: Online self-help intervention

SUMMARY:
This is a study on internet-based self-help for stress related to the COVID-19 pandemic. College and university students who score in the moderate or higher range on a stress measure during the COVID-19 pandemic will be invited to participate in this study. Participants will be randomly assigned to receive access to an internet-based self-help program for stress resilience and coping with the COVID-19 pandemic or care as usual. Stress and psychosocial symptoms will be assessed via questionnaire at baseline (pre-randomization), one month post-randomization, and three months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or higher stress as assessed using Stress subscale of the Depression Anxiety Stress Scales-Short Form
* Current student at a college or university in the United States
* Able to provide consent
* Proficient in English

Exclusion Criteria:

* Below age 18
* Failure to meet any of above inclusion criteria
* Current participant in separate randomized controlled trial being conducted by this research group examining efficacy of SilverCloud Health interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in stress | Measured at baseline, one month, and three months. The primary outcome is change in scale scores from baseline to one month. Change from baseline to three months will also be examined as a secondary outcome.
  Stress assessed using the Stress subscale of the Depression, Anxiety, Stress Scales-Short Form (7 of 21 items; self-report; possible range = 0-42)

SECONDARY OUTCOMES:
Change in anxiety | Measured at baseline, one month, and three months. Outcomes include change in scale score from baseline to one month and change in scale score from baseline to three months.
  Anxiety assessed using the Anxiety subscale of the Depression, Anxiety, Stress Scales-Short Form (7 of 21 items; self-report; possible range = 0-42)
Change in depression | Measured at baseline, one month, and three months. Outcomes include change in scale score from baseline to one month and change in scale score from baseline to three months.
  Depression assessed using the Depression subscale of the Depression, Anxiety, Stress Scales-Short Form (7 of 21 items; self-report; possible range = 0-42)
Change in perceived stress | Measured at baseline, one month, and three months. Outcomes include change in scale score from baseline to one month and change in scale score from baseline to three months.
  Perceived stress assessed using the Perceived Stress Scale-10 (10 items, self-report; possible range = 0-40)
Change in coronavirus-related stress | Measured at baseline, one month, and three months. Outcomes include change in subscale scores from baseline to one month and change in subscale scores from baseline to three months.
  Coronavirus-related stress assessed using the COVID Stress Scales (6-item self-report subscales assessing the following forms of coronavirus-related stress: danger, socioeconomic consequences, xenophobia, contamination fears, traumatic stress, compulsive checking; subscale scores range from 0 to 24)

OTHER OUTCOMES:
Change in screening status for major depressive disorder | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for major depressive disorder using the Patient Health Questionnaire-9 (9 items, self-report, possible range = 0-40, probable depression indicated by score of 10 or higher)
Change in screening status for generalized anxiety disorder | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for generalized anxiety disorder using the Generalized Anxiety Disorder Questionnaire-IV (9 items, self-report, probable generalized anxiety disorder indicated if participants endorse all diagnostic criteria)
Change in screening status for social anxiety disorder | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for social anxiety disorder using the Social Phobia Diagnostic Questionnaire (25 items, self-report; probable social anxiety disorder indicated if participants endorse all diagnostic criteria)
Change in screening status for panic disorder | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for panic disorder using Panic Disorder Self-Report (24 items, self-report, probable panic disorder indicated if participants endorse all diagnostic criteria)
Change in screening status for anorexia nervosa | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for anorexia nervosa using Stanford-Washington University Eating Disorder scale (14 items, self-report; probable anorexia nervosa indicated if participants score 59 or higher (out of 100) on weight concerns items and endorse current body mass index ≤ 18.45)
Change in screening status for bulimia nervosa/binge eating disorder | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for bulimia nervosa or binge eating disorder using Stanford-Washington University Eating Disorder scale (14 items, self-report; probable bulimia nervosa or binge eating disorder indicated if participants do not screen positive for probable anorexia nervosa and endorse six or more instances of binge-eating, self-induced vomiting, or diuretic or laxative misuse in the past three months).
Change in screening status for insomnia | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for insomnia using Insomnia Severity Index (7 items, self-report, scores range from 0 to 28; probable insomnia indicated by score of 15 or higher).
Change in screening status for alcohol use disorder | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for alcohol use disorder using Alcohol Use Disorders Identification Test-C (3 items, self-report, scores range from 0 to 12; probable alcohol use disorder indicated by score of 4 or higher for males and 3 or higher for females).
Change in screening status for posttraumatic stress disorder | Measured at baseline, one month, and three months. Outcomes include change in screening status from baseline to one month and change in screening status from baseline to three months.
  Screening for posttraumatic stress disorder using Primary Care PTSD Screen (4 items, self-report, scores range from 0 to 4; probable posttraumatic stress disorder indicated by score of 3 or higher).

CONTACTS AND LOCATIONS:
Overall Officials: Gavin N Rackoff, MS, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rackoff GN, Fitzsimmons-Craft EE, Taylor CB, Eisenberg D, Wilfley DE, Newman MG. A Randomized Controlled Trial of Internet-Based Self-Help for Stress During the COVID-19 Pandemic. J Adolesc Health. 2022 Aug;71(2):157-163. doi: 10.1016/j.jadohealth.2022.01.227. Epub 2022 Feb 4. PMID 35351353